CLINICAL TRIAL: NCT01255982
Title: Functional Assessment of Patients With Acute Bipolar Depression After 8 Months of Follow-up
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NES-DUM-2010/1
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: Bipolar depression; subsyndromal symptoms; functioning; cognitive function
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Diagnosed with bipolar I or II disorder, and with an acute episode of bipolar depression at inclusion

SUMMARY:
This study aims to study prospectively for 8 months a sample of bipolar patients with acute depressive episode in order to identify that factors associated with functional impairment, with especial attention to the presence of subsyndromal symptoms beyond the acute phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder I or II (DSM-IV-TR)
* Acute depressive episode at inclusion

Exclusion Criteria:

* Inability (in investigator´s opinion) to carry out the follow-up plan
* Patients participating or having participated within previous 6 months, in clinical trials
* Mental retardation or any other medical condition affecting cognitive performance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Outpatients from Mental Health Centres or Psychiatric Offices, diagnosed with bipolar I or II disorder experiencing an acute depressive episode.
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Difference between basal and final Functional Assessment Staging (FAST) score to evaluate the functional change | Range of Days 0-3

SECONDARY OUTCOMES:
FAST score to estimate the proportion of patients that not achieve functional remission | Range of Days 0-3
Test Screen for Cognitive Impairment in Psychiatry (SCIP) to evaluate cognitive impairment both in the depressive phase and during clinical remission | Range of Days 0-3
Mood chart (self-report) | Range of Days 0-3
The presence of subsyndromal symptoms after the acute depressive phase using Montgomery-Asberg Depression Rating Scale (MADRS), Young Mania Rating Scale (YMRS), Diagnostic and Statistical Manual of Mental disorders (DSM-IV-TR) | Range of Days 0-3

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - Research Site, Elche, Alicante
  - Research Site, Villajoyosa, Alicante
  - Research Site, Almería, Almería
  - Research Site, Barcelona, Barcelona
  - Research Site, Granollers, Barcelona
  - Research Site, San Boit de LLobregat, Barcelona
  - Research Site, Córdoba, Cordoba
  - Research Site, Granada, Granada
  - Research Site, Lleida, Lerida
  - Research Site, Monforte de Lemos, Lugo
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Tudela, Navarre
  - Research Site, Ourense, Orense
  - Research Site, Palencia, Palencia
  - Research Site, Palma de Mallorca, Palma de Mallorca
  - Research Site, Mos, Pontevedra
  - Research Site, Langreo, Principality of Asturias
  - Research Site, Seville, Sevilla
  - Research Site, Tarragona, Tarragona
  - Research Site, Catarroja, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Zamora, Zamora
  - Research Site, Zaragoza, Zaragoza